CLINICAL TRIAL: NCT01782209
Title: Natural History of Infection Caused by BK Virus (and Other Opportunistic Viral Pathogens) in Renal Transplant Recipients
Brief Title: BK Virus Infection (Viremia) Natural History in Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Richard J Whitley, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: DMID 11-0071
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: BK Virus (BKV) Viremia
Keywords: BK virus viremia; renal transplant; other viral pathogens
MeSH Terms: conditions — Viremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be processed for serum and then evaluated for BK virus DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study is to establish the natural history of BK virus viremia and other possible opportunistic viral pathogens in renal transplants recipients.

DETAILED DESCRIPTION:
This is a Natural History study in renal or renal-pancreas transplant recipients. In an effort to capture patients early in the course of an evolving BK virus infection and avoid patients who have already developed evidence of BKV-induced nephropathy (BKVN), this protocol will emphasize the initiation of screening in the early post-transplant period. Patients who have undergone renal or renal/pancreas transplantation within 4 weeks, but not more than 90 day previously, will be asked to participate and then consented to be enrolled in a Natural History-Surveillance period for up to approximately 24 months. Participants enrolled in this study will provide valuable natural history data regarding BKV viremia, and potentially other viral pathogen, in the post-renal transplant period. Participants will provide blood samples to undergo measurement for plasma BKV DNA by PCR approximately every 6 weeks, to be resulted in real time at the UAB Diagnostic Virology Laboratory at UAB.

ELIGIBILITY:
Inclusion Criteria:

Renal or renal-pancreas transplant patients who are within 4 weeks and not more than 90 days post-transplant with or without qualifying BKV viremia Age greater than or equal to 18 years; Provides written informed consent.

Exclusion Criteria:

Evidence of proven or suspected BKVN by clinical or pathologic diagnostic criteria Loss of renal graft function Initiation of chronic dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female renal or renal-pancreas transplant recipients ages 18 and older at risk for BKV infection
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Whitley, MD, Principal Investigator — University of Birmingham at Alabama; John W Gnann, MD, Study Chair — Medical University of South Carolina
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado at Denver and HSC, Denver, Colorado
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, Barnes Jewish Hospital, St Louis, Missouri
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Renal Transplant Patients: Male and female renal or renal-pancreas transplant recipients at risk for BK virus infection
Period: Overall Study
Arm/Group | Renal Transplant Patients
Started | 335
Completed | 225
Not Completed | 110

BASELINE CHARACTERISTICS:
Arm/Group | Renal Transplant Patients
Number analyzed (Participants) | 335
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 313
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 100
  White | 214
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 335

OUTCOME MEASURES:

1. Primary Outcome: Incidence of BKV Viremia in the Study Population of Screened Renal or Renal-pancreas Transplant Subjects
Description: We will measure the number of subjects screened who develops BK viremia within 4 weeks and up to 24 months after renal transplant
Time Frame: within 4 weeks and up to 24 months after renal transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Transplant Patients
Number analyzed (Participants) | 335
Participants | 58
Statistical Analysis 1: Comparison: Renal Transplant Patients; Test type: Other; Incidence = 17.3, 95% CI 2-sided [13.4 to 21.8] — 95% Clopper-Pearson Confidence Interval

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Renal Transplant Patients
All-Cause Mortality (participants affected / at risk) | 4/335
Serious Adverse Events (participants affected / at risk) | 0/335
Other Adverse Events (participants affected / at risk) | 1/335
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Transplant Patients (N=335)
Bruising on left arm (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT01782209/Prot_SAP_000.pdf